CLINICAL TRIAL: NCT05367401
Title: A Phase Ib/II, Open Label, Proof-of-concept Study of Sabatolimab and Magrolimab-based Therapy for Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: A Study of Sabatolimab and Magrolimab-based Treatment in AML or Higher Risk MDS Participants
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: waiting for update from Study Lead
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453B12205; 2021-003263-10 (EudraCT Number)
Record Dates: First submitted 2022-04-21; First posted 2022-05-10 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
Keywords: relapsed/refractory; R/R; Phase 1/2; Sabatolimab; Magrolimab; Azacitidine; Myelodysplastic Syndromes; MDS; Acute myeloid leukemia; AML; TIM-3; CD47
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Recurrence | interventions — sabatolimab; magrolimab; Azacitidine

STUDY DESIGN:
Intervention Model Description: Safety run in (1L higher risk MDS + 1L unfit AML) followed by parallel expansion cohorts (1L higher risk MDS, 1L unfit AML, relapsed/refractory AML)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1L higher risk MDS (Experimental): Participants with 1L MDS will receive sabatolimab and magrolimab in combination with azacitidine
  Interventions: Drug: Sabatolimab; Drug: Magrolimab; Drug: Azacitidine
- 1L unfit AML (Experimental): Participants with 1L AML unfit for intensive chemotherapy will receive sabatolimab and magrolimab in combination with azacitidine
  Interventions: Drug: Sabatolimab; Drug: Magrolimab; Drug: Azacitidine
- Relapsed/refractory AML previously treated with venetoclax and azacitidine (Experimental): Participant with relapsed/refractory AML will receive sabatolimab and magrolimab (in absence of complete response (CR), Complete Remission with incomplete hematologic recovery (CRi) or Morphologic Leukemia-Free State (MLFS) after 2 cycles, participants will be allowed to also receive azacitidine)
  Interventions: Drug: Sabatolimab; Drug: Magrolimab

INTERVENTIONS:
Drug: Sabatolimab — Solution for intravenous infusion
  Other Names: MBG453
Drug: Magrolimab — Solution for intravenous infusion
  Other Names: GS-4721
Drug: Azacitidine — Solution for subcutaneous injection or intravenous infusion
  Arms: 1L higher risk MDS; 1L unfit AML

SUMMARY:
This study is to determine the safety and preliminary efficacy of sabatolimab in combination with magrolimab and azacitidine in adult participants with 1L unfit Acute Myeloid Leukemia (AML) or with 1L higher risk Myelodysplastic Syndromes (MDS), and sabatolimab in combination with magrolimab in participants with relapsed or refractory (R/R) AML.

DETAILED DESCRIPTION:
The primary purpose of the Safety run-in is to rule out excessive toxicity and investigate safety of the combination of sabatolimab with azacitidine and magrolimab in previously untreated participants with higher-risk MDS and unfit AML. The primary purpose of the combined Safety Run-in and Expansion is to assess the preliminary efficacy of the combination of sabatolimab with magrolimab with (cohort 1 and 2) or without (cohort 3) azacitidine in terms of achieving complete remission in 3 different indications:

* Previously untreated participants with AML, who are unfit for intensive chemotherapy (1L unfit AML - cohort 1),
* Previously untreated participants with higher-risk MDS (1L higher risk MDS - cohort 2),
* Participants with R/R AML after having been previously treated with only first line venetoclax in combination with hypomethylating agent (VEN+HMA) (R/R AML - cohort 3).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Age ≥ 18 years at the date of signing the informed consent form (ICF)
3. Newly diagnosed with AML based on 2016 WHO classification (Arber et al 2016) and not suitable for intensive chemotherapy defined as: age ≥75, ECOG performance Status 2 or 3, or any of the following comorbidities: severe cardiac comorbidity (including congestive heart failure, LVEF ≤ 50%, chronic stable Angina) , pulmonary comorbidity (DLCO ≤ 65% or FEVI ≤ 65%). moderate hepatic impairment (with total Bilirubin >1.5 to 3x ULN) , renal impairment (eGFR≥ 30 ml/min/1.73m^2 to 45 30 ml/min/1.73m^2), or other comorbidity incompatible with intensive chemotherapy per Investigator assessment and approved by the Novartis Medical monitor) OR

   Morphologically confirmed diagnosis of myelodysplastic syndrome (MDS) based on 2016 WHO classification (Arber et al 2016), that is intermediate, high or very high risk (higher risk) based on the revised International Prognostic Scoring System (IPSS-R) (Greenberg et al 2012), previously untreated for higher risk MDS [1L higher risk MDS]:
   * Intermediate (>3-4.5 points)
   * High (> 4.5-6 points)
   * Very high (> 6 points) OR (for expansion only) Participants with AML relapsed or refractory to venetoclax in combination with a hypomethylating agent (VEN+HMA) as defined by failure to achieve bone marrow blast <5% after at least 2 cycles of VEN+HMA (refractory) or relapsed after having achieved BM blast <5% following previous treatment with VEN+HMA as first and the only line of treatment for AML
4. Eastern Cooperative Oncology Group (ECOG) performance status must be 0-2 for participants ≥ 75 years of age, OR 0-3 for participants < 75 years of age
5. White blood cell (WBC) count ≤ 20 x 10^3/μL prior to first dose of study treatment (may be reduced with leukapheresis, hydroxyurea, or oral etoposide)
6. Hemoglobin ≥ 9 g/dL prior to initial dose of study treatment. Transfusions are allowed to meet hemoglobin eligibility prior to first dose of study treatment

Exclusion Criteria:

1. Prior treatment with CD47 or signal regulatory protein alpha (SIRPα) targeting agents
2. Prior exposure to TIM-3 directed therapy
3. Prior therapy with immune checkpoint inhibitors (eg, anti-CTLA4, anti-PD-1, anti-PDL1, or anti-PD-L2) or cancer vaccines is not allowed if the last dose of the drug was administered within 4 months prior to start of the study treatment
4. For participants with higher risk MDS only: Previous first-line treatment for intermediate, high, very high risk (higher risk) MDS (based on IPSS-R) with any antineoplastic agents including for example chemotherapy and hypomethylating agents such as decitabine or azacitidine.

   For participants with newly diagnosed AML only: Previous treatment at any time, with any approved or investigational antineoplastic agents for AML or higher risk MDS.

   Prior and concurrent therapy with hydroxyurea or oral etoposide (to reduce WBC count), supportive care ruxolitinib, erythroid and/or myeloid growth factors are allowed.
5. Acute promyelocytic leukemia
6. Known inherited or acquired bleeding disorders
7. Patients with CNS leukemia or neurologic signs and symptoms suggestive of CNS leukemia (unless CNS leukemia had been excluded)

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2029-10-26 (Estimated); Study Completion 2029-10-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with dose limiting toxicities (only for participants enrolled in the safety run-in part) | Cycle 1 Day 1 to the end of Cycle 2 (up to 14 days from the planned cycle 3 Day 1) ; Cycle = 28 Days
  Assessment of tolerability of sabatolimab and magrolimab given together with azacitidine
Percentage of participants achieving complete remission (CR) according to Investigator assessment per treatment arm | Up to 4 years from last patient first treatment
  Assessing the Complete Remission (CR) Rate in each treatment arm (including participants from safety run-in and expansion) per IWG -Cheson 2003 and ELN AML recommendations - Doehner 2017 (AML) and per modified IWG-MDS criteria- Cheson 2006 (MDS) in each treatment arm.

SECONDARY OUTCOMES:
Anti-drug-antibody prevalence at baseline | prior to first dose of sabatolimab on week 2 Day 1 and first dose of magrolimab on week 1 day 1
  Measuring immunogenicity to sabatolimab and magrolimab prior to exposure
Anti-drug-antibody prevalence on treatment | Throughout study until 90 day safety follow up for sabatolimab and 30 day safety follow up for magrolimab
  Measuring immunogenicity to sabatolimab and magrolimab on treatment and after treatment
Peak of Serum Concentration (Cmax) sabatolimab and magrolimab | Day 1 of week 2, 5, 13 for sabatolimab. Day 1 or week 1, 5, 13 for magrolimab
  Maximal serum concentration of sabatolimab and magrolimab
Trough serum concentration (Cmin) sabatolimab | Day 1 of week 2, 5, 9, 13, 25, 37, 49, 73, 97, end of treatment (EOT) (within 7 days after the last dose of study treatment), 30 days after last dose of sabatolimab, and 90 days after the last dose of sabatolimab for sabatolimab
  Concentration of sabatolimab prior to next dosing or after end of treatment
Trough serum concentration (Cmin) magrolimab | Day 1 or week 1, 2, 5, 9, 13, 25, 37, 49, 73, 97, end of treatment (EOT) (within 7 days after the last dose of study treatment), 30 days after last dose of magrolimab for magrolimab
  Concentration of magrolimab prior to next dosing or after end of treatment
Time from first occurrence of CR (complete remission) to relapse from CR or death due to any cause whichever occurs first (All 3 arms) | Up to 4 years from last patient first treatment
  Assessing the duration of complete response defined as time from first occurence of CR per IWG -Cheson 2003) and ELN Doehner 2017 AML recommendations (AML) and per modified IWG-MDS criteria (MDS) to relapse from CR per IWG CHeson 2003 and ELN -Doehner 2017 AML recommendations (AML) and per modified IWG-MDS criteria Cheson 2006 (MDS) or death due to any cause ,whichever occurs first
Percentage of participants achieving CR, CR with incomplete hematologic recovery (CRi), or partial response (PR) as per Investigator (1L unfit AML and R/R AML arms only) | Up to 4 years from last patient first treatment
  Assessing the overall response rate defined as proportion of participants achieving CR, CR with incomplete hematologic recovery (CRi), or partial response (PR) as per investigator assessment as per ELN -Doehner 2017 and IWG criteria -Cheson 2003
Percentage of participants achieving CR or CRi (1L unfit AML and R/R AML arms only) | Up to 4 years from last patient first treatment
  Assessing the [CR + CRi] rate defined as proportion of patients achieving complete remission or complete remission with incomplete hematologic recovery per IWG - Cheson 2003 and ELN AML recommendations -Doehner 2017 (AML)
Percentage of participants achieving CR or CRh (1L unfit AML and R/R AML arms only) | Up to 4 years from last patient first treatment
  Assessing the [CR + CR with partial hematologic recovery (CRh)] rate defined as proportion of patients achieving complete remission or complete remission with partial hematological recovery per IWG and ELN AML recommendations (AML)
Percentage of participants achieving CR with Measurable Residual Disease (MRD)-negative status(1L unfit AML and R/R AML arms only) | Up to Day 1 of cycle 13 ; Cycle=28 days
  Assessing the rate of MRD-negative CR participants defined as proportion of participants in complete remission with no detectable minimal residual disease
Percentage of participants achieving CR or CRi with MRD-negative status (1L unfit AML and R/R AML arms only) | Up to Day 1 of Cycle 13 ; Cycle =28 days
  Rate of MRD-negative participants Assessing the rate of MRD-negative CR /CRi participants defined as proportion of participants in either complete remission or complete remission with incomplete hematologic recovery with no detectable minimal residual disease
Percentage of participants achieving CR, marrow CR (mCR), partial response (PR), hematologic improvement (HI) per Investigator assessment (1L higher risk MDS arm only) | Up to 4 years from last patient first treatment
  Assessing the overall response rate defined as proportion of patients achieving CR, marrow CR (mCR), partial response (PR), hematologic improvement (HI) per Investigator assessment according to modified IWG-MDS response criteria- Cheson 2006
Percentage of participants who are red blood cells (RBC)/platelets transfusion independent (1L MDS arm only) | From start of treatment up to until 4 years after last patient first treatment
  Assessing the improvement in RBC/platelets transfusion independence
Duration of transfusion independence (1L MDS arm only) | From start of treatment up to until 4 years after last patient first treatment
  Assessing the time to RBC/platelets transfusion independence

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The Trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com